CLINICAL TRIAL: NCT00003404
Title: A Prospective Study of Adjuvant Radiation Therapy After Resection of Borderline and Malignant Phyllodes Tumors
Brief Title: Radiation Therapy After Surgery in Treating Women With Phyllodes Tumor of the Breast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Richard J. Barth,Jr., Chief, Section of General Surgery, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9801 CDR0000066410; P30CA023108 (NIH); DMS-9801; DMS-12752; NCI-V98-1442
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; phyllodes tumor
MeSH Terms: conditions — Breast Neoplasms; Phyllodes Tumor | interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Adjuvant Radiotherapy (Experimental): Adjuvant radiation was started within 12 weeks of local excision or breast re-excision.
  Interventions: Radiation: Adjuvant Radiotherapy

INTERVENTIONS:
Radiation: Adjuvant Radiotherapy — Adjuvant radiation therapy

SUMMARY:
PURPOSE: This phase II trial studied how well radiation therapy works after surgery in treating women with phyllodes tumor of the breast.

RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Radiation therapy following surgery may be effective in treating patients with phyllodes tumor of the breast.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the local recurrence rate in women with phyllodes tumors of the breast previously treated with local excision with negative margins and are now treated with adjuvant radiotherapy.
* Determine the survival rate in patients treated with this regimen.

METHODS: Within 12 weeks after prior local excision or breast reexcision, patients underwent adjuvant radiotherapy 5 days a week for a total of 28 treatments. Patients were then followed every 6 months for 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

1. Histologically proven phyllodes tumors of the breast with borderline or malignant grade, defined as 1 of the following:

   1. Borderline, defined as 5-9 mitoses/10 high power fields (HPF), pushing or infiltrating margins, 2+ atypia
   2. Malignant, defined as 10 or more mitoses/10 HPF, predominantly infiltrating margins, usually 3+ atypia with occasional 2+ atypia
2. Must have been excised with breast-conserving resection and no positive margins
3. Local recurrence of a previously excised phyllodes tumor allowed if the recurrence is in the area of the prior excision
4. No prior breast carcinoma or ductal carcinoma in situ in the ipsilateral breast
5. Hormone receptor status: Not specified

PATIENT CHARACTERISTICS:

1. Age: 18 and over
2. Sex: Female
3. Menopausal status: Not specified
4. Performance status: Not specified
5. Life expectancy: Not specified
6. Hematopoietic: Not specified
7. Hepatic: Not specified
8. Renal: Not specified
9. Other:

   1. Not pregnant
   2. Negative pregnancy test
   3. Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

1. Biologic therapy: Not specified
2. Chemotherapy: Not specified
3. Endocrine therapy: Not specified
4. Radiotherapy: No prior radiotherapy to the ipsilateral breast
5. Surgery: See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1998-01 (Actual); Primary Completion 2008-11-17 (Actual); Study Completion 2008-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Barth, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Result] Barth RJ Jr, Wells WA, Mitchell SE, Cole BF. A prospective, multi-institutional study of adjuvant radiotherapy after resection of malignant phyllodes tumors. Ann Surg Oncol. 2009 Aug;16(8):2288-94. doi: 10.1245/s10434-009-0489-2. Epub 2009 May 8. PMID 19424757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from a total of 30 different institutions. Half of the patients were treated at community-based treatment centers, and half were treated at academic medical centers.
Period: Overall Study
Arm/Group | Adjuvant Radiotherapy
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adjuvant Radiotherapy
Number analyzed (Participants) | 46
Age, Continuous [Mean (Full Range); unit: years] | 49 [18 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Local Recurrence Rate
Description: Local recurrence rate of phyllodes tumors
Time Frame: 36 months after initial excision
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Radiotherapy
Number analyzed (Participants) | 46
Participants | 0
Statistical Analysis 1: Comparison: Adjuvant Radiotherapy; Test type: Other; rate of occurance = 0.35, 95% CI 2-sided [0 to 8] — The local recurrence rate was estimated by dividing the number of recurrences by the total sample size. An exact 95% confidence interval (95% CI) for this rate was determined by binomial distribution

2. Secondary Outcome: Survival Rate
Description: Survival will be tracked for 10 years after initial resection of first participant treated.
Time Frame: Approximately 5 years
Population: All patients received adjuvant radiotherapy as specified in the protocol. No patients were lost to follow-up. Duration of follow-up ranged from 12 to 129 months, with a median follow-up of 56 months and a mean follow-up of 60 months. Ninety percent of the patients were followed for at least 2 years.
Measure: Count of Participants; unit: Participants
Groups:
- Adjuvant Radiotherapy: Adjuvant radiation after local excision or breast re-excision.
Arm/Group | Adjuvant Radiotherapy
Number analyzed (Participants) | 46
Participants | 2

ADVERSE EVENTS:
Arm/Group | Adjuvant Radiotherapy
All-Cause Mortality (participants affected / at risk) | 2/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No